CLINICAL TRIAL: NCT02481531
Title: Growth and Tolerance of Cow's Milk-Based Infant Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3387-1
Record Dates: First submitted 2015-06-19; First posted 2015-06-25 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Previously marketed infant formula (Active Comparator): Cow's milk-based infant formula
  Interventions: Other: Previously marketed infant formula
- Previously marketed formula using a similar protein (Experimental): Cow's milk-based infant formula
  Interventions: Other: Previously marketed formula using a similar protein

INTERVENTIONS:
Other: Previously marketed infant formula
  Arms: Previously marketed infant formula
Other: Previously marketed formula using a similar protein
  Arms: Previously marketed formula using a similar protein

SUMMARY:
This clinical trial will evaluate the growth, tolerance, and iron status of infants who consume an investigational infant formula containing a nutrient-rich whey protein compared to a previously marketed infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 10-14 days of age at randomization
* Term infant with birth weight of a minimum of 2500 grams
* Solely formula fed
* Signed Informed Consent and Protected Health Information

Exclusion Criteria:

* Anemia at time of birth
* Current use of iron or iron-containing supplements
* History of underlying metabolic or chronic disease or immunocompromised
* Feeding difficulties or formula intolerance

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 373 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Body weight measured at each study visit | 12 months
  Measurement collected with a calibrated infant scale

SECONDARY OUTCOMES:
Body length measured at each study visit | 12 months
  Measurement collected with a standardized length board
Head circumference measured at each study visit | 12 months
  Measurement collected with a standardized measuring tape
Parental recall of study formula intake at each study visit | 12 months
Parental recall of stool consistency measured at each study visit | 12 months
Blood Collection | Once at 12 months
  Composite measure of hemoglobin, hematocrit, ferritin, and c-reactive protein
Medically-confirmed adverse events collected throughout the study period | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wu, M.D., Study Director — Mead Johnson and Company
Locations (22):
- United States (22):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Pediatrics East - Alabama Clinical Therapeutics, Pinson, Alabama
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Norwich Pediatric Group, P.C., Norwich, Connecticut
  - Children's Research, LLC, Altamonte Springs, Florida
  - Deaconess Clinical Research, Evansville, Indiana
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatrics/Adult Research, Bardstown, Kentucky
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Woburn Pediatic Associates, Woburn, Massachusetts
  - Pediatric Associates of Mt. Carmel, Inc, Cincinnati, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - UHMP Comprehensive Pediatrics, Westlake, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - The Jackson Clinic - North Jackson, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - DCOL Center for Clinical Research, Longview, Texas

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831